CLINICAL TRIAL: NCT07347379
Title: Long-Term Clinical Outcomes Of Subjects Enrolled In The RxSight Light Adjustable Lens (LAL) And Light Delivery Device (LDD) New Enrollment Study
Status: Enrolling by invitation | Type: Observational
Sponsor: RxSight, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CSP-1003
Record Dates: First submitted 2025-12-04; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Aphakia Cataract
Keywords: Light Adjustable Lens LAL Intraocular lens

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Light adjustable lens (LAL) and Light Delivery Device (LDD): Light adjustable lens (LAL) and Light Delivery Device (LDD)
  Interventions: Device: Light Adjustable lens (LAL) and Light Delivery Device (LDD)
- Control IOL: Control IOL
  Interventions: Device: Control IOL

INTERVENTIONS:
Device: Light Adjustable lens (LAL) and Light Delivery Device (LDD) — Experimental treatment group received Light adjustable lens with Light delivery Device treatments
  Groups: Light adjustable lens (LAL) and Light Delivery Device (LDD)
Device: Control IOL — Control treatment group received a Control IOL
  Groups: Control IOL

SUMMARY:
This is an observational, follow up study of subjects previously enrolled in the "RxSight Light Adjustable Lens (LAL) and Light Delivery Device (LDD) New Enrollment Study". The primary objective of this study is to collect long-term safety and effectiveness data on RxSight LAL and Control IOL in subjects previously implanted in the "RxSight Light Adjustable Lens (LAL) and Light Delivery Device (LDD) New Enrollment Study".

ELIGIBILITY:
Inclusion Criteria:

* Subject and study eye with prior participation in the CSP-029 study.

Exclusion Criteria:

* Subjects with serious co-morbid conditions that in the judgment of the investigator makes inclusion in the study not in the best interest of the subject.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include up to 500 subjects who previously participated in the CSP-029 study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Mean absolute manifest refraction spherical equivalent (|MRSE|) at the Long-Term follow up visit compared between the RxSight LAL and Control group | Up to 55 months
Mean manifest cylinder at the Long-Term follow up visit compared between the RxSight LAL and Control group | Up to 55 months

CONTACTS AND LOCATIONS:
Locations (1):
- Focal Point Vision, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No